CLINICAL TRIAL: NCT03762187
Title: Effects of a Brief Affirmation Intervention on HIV-related Distress and Positive Living Intentions Among Individuals Recently Diagnosed With HIV in Lesotho
Brief Title: A Brief Affirmation Intervention on HIV-related Distress and Positive Living in Lesotho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Santa Barbara (Other)
Collaborators: Fulbright (Other); Ministry of Health, Lesotho (Other Government)
Responsible Party: Principal Investigator, David Sherman, Professor, University of California, Santa Barbara
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0333
Record Dates: First submitted 2018-11-01; First posted 2018-12-03 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Self-affirmation Plus Positive Living Counseling; Counseling

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of the two conditions.
Who Masked: Participant, Care Provider
Masking Description: Neither patients nor counselors were aware of participants' assigned condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-affirmation (Experimental): Participants completed a written self-affirmation manipulation before completing the standard counseling provided by the clinic.
  Interventions: Behavioral: Self-affirmation; Behavioral: Positive living counseling
- Positive living counseling (Active Comparator): Participants completed the standard counseling provided by the clinic (treatment as usual control condition).
  Interventions: Behavioral: Positive living counseling

INTERVENTIONS:
Behavioral: Self-affirmation — Individuals select important values and then write about why that value is important to them.
  Arms: Self-affirmation
Behavioral: Positive living counseling — Each of the clinics from which participants were recruited conducts positive living counseling as part of their treatment programs. This counseling is conducted by counselors who are trained and monitored by the Lesotho Network of AIDS Support Organizations (LENASO) and consistent with the positive prevention framework (see Bunnell et al., 2005 for description). Each counseling session focused on addressing positive living goals such as the importance of taking one's medications on time and every day, using protection with every partner, and the importance of maintaining a healthy lifestyle.

SUMMARY:
This study is interested in the stress associated with being HIV positive and looking at ways to reduce that stress. Individuals who are HIV positive face a number of nontrivial threats and stressors: the burden of illness, loss of work, stigmatization, and the chance of death. The study investigates the use of self-affirmation to reduce some of these threats and stressors. Self-affirmation may helping people to cope with these threats and stressors by reminding individuals of other valued aspects of themselves, thus reducing the impact, both psychologically and physiologically, of these threats. Experimentally induced affirmations in which individuals are asked to write about values that are important to the self have been shown to reduce physiological stress among healthy student populations (Sherman, Bunyan, Creswell, & Jaremka, 2009).

This research will be conducted in collaboration with the global health organizations, PSI who is already providing counseling to those living with HIV on how to reduce the spread of HIV and how to live a healthy life with HIV. These counseling sessions take place at local clinics and hospitals while individuals are waiting to be seen for treatment and are completely voluntary.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* A CD4 count of less than or equal to 500 cells/mm3 or have significant symptomatology and HIV co-illness (WHO HIV clinical stage 3 or 4) to be eligible to start antiretroviral therapy

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Post-intervention survey conducted immediately after intervention session
  Participants were asked to complete an abbreviated version of the Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983), a well validated measure of participants' current stress. For this scale, participants are asked to rate their agreement with statements such as "Today, I feel nervous and stressed" or "Today I feel that difficulties are piling up so high that I cannot overcome them" using a 6-point Likert scale anchored from 1= "Very Much Disagree" to 6 = "Very Much Agree".
Intrusion subscale of impact of events scale | Post-intervention survey conducted immediately after intervention session
  Participants completed questions regarding their current experience of intrusive thoughts related to HIV adapted from the intrusion subscale of the Impact of Events Scale (Horowitz, Wilner, & Alvarez, 1979). This measure was designed to assess distress caused by traumatic events. The impact of events scale is a well-validated measure that is often used (in combination with the DSM-IV) to assess post-traumatic stress disorder. In essence, this measure was designed to assess how traumatized participants felt by their HIV diagnosis. Participants rated their agreement with statements such as "Today, any reminder of HIV brings back feelings about it" and "Today, I think about HIV even when I don't mean to" using a 1= "Very Much Disagree" to 6 = "Very Much Agree" scale.
Concerns about dying | Post-intervention survey conducted immediately after intervention session
  Participants indicated to what extent they were currently concerned about dying using a single item, "Today, I find myself worrying about dying". Participants indicated their agreement with that statement using a 6-point Likert scale from 1= "Very Much Disagree" to 6 = "Very Much Agree", with higher numbers indicating greater worries about dying.
Distressing emotions related to HIV | Post-intervention survey conducted immediately after intervention session
  Participants indicated to what extent they were experiencing distressing emotions related to HIV on a 5-point Likert scale from 1="Never" to 5="Always", with higher numbers indicating a greater frequency of distressing emotions related to HIV.
Future behavioral intentions | Post-intervention survey conducted immediately after intervention session
  Participants were asked to rate their agreement with statements regarding their future intentions to engage in positive living behaviors using a 6-point Likert scale from from 1= "Very Much Disagree" to 6 = "Very Much Agree". In particular, participants were asked to indicate their intention to use condoms in the future by indicating their agreement with statements such as, "If a sexual partner didn't want to use condoms, we would have sex without using condoms" or "It is a hassle to use condoms". Participants indicated their intention to take their medications by indicating their agreement with the statements, "I will take my medication regularly" and "I have trouble taking my medication as I am supposed to (reversed)". Additionally, participants indicated their intention to have non-concurrent sexual partners using the statement "I will only have one sexual relationship at a time".

SECONDARY OUTCOMES:
Physical health measures | Post-intervention survey conducted immediately after intervention session
  In order to assess participants' baseline self-reported health, participants completed the general health subscale of the RAND 36-item Short Form Health Survey, a well-validated measure designed to assess health that is utilized by many health organizations, including Medicare, to assess and monitor healthcare outcomes. Participants were asked to answer five questions regarding their current health using a 5-point Likert scale.

IPD SHARING:
Plan to Share IPD: No